CLINICAL TRIAL: NCT04646746
Title: HIAMBA-1 - the Effects of Nude Barley and Gene-modified High-amylose Barley on Postprandial Glucose Metabolism in Subjects With Type 2 Diabetes
Brief Title: Acute Studies on the Glycemic Index After Intake of Different Sorts of Barley in Subjects With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Innovation Fund Denmark (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: HIAMBA-1
Record Dates: First submitted 2020-11-16; First posted 2020-11-30 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes
Keywords: Glycemic index; Postprandial; Barley
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Flour

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, cross-over, acute, dietary intervention study
Who Masked: Participant, Investigator
Masking Description: Color labeling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 100 g of 100% wheat bread (Experimental): Intake of 250 ml of tap water and 100 g of bread baked with 100% wheat flour (regular commercial available wheat flour). Consumed over maximum 10 minutes at time 0 min after overnight fasting. At one of four visits.
  Interventions: Dietary Supplement: 100% wheat
- Nude barley 50% (Experimental): Intake of 250 ml of tap water and 100 g of bread baked with 50% nude barley flour and 50% wheat flour. Consumed over maximum 10 minutes at time 0 min after overnight fasting. At one of four visits.
  Ancient nude barley naturally bred in corporation with PlantCarb ApS and researchers at Aarhus and Copenhagen Universities. The wheat flour is standard commercial available flour.
  Interventions: Dietary Supplement: 50% nude barley and 50% wheat
- Nude barley 75% (Experimental): Intake of 250 ml of tapwater and 100 g of bread baked with 75% nude barley flour and 25% wheat flour. Consumed over maximum 10 minutes at time 0 min after overnight fasting. At one of four visits.
  Ancient nude barley naturally bred in corporation with PlantCarb ApS and researchers at Aarhus and Copenhagen Universities. The wheat flour is standard commercial available flour.
  Interventions: Dietary Supplement: 75% nude barley and 25% wheat
- Gen-modified high-amylose barley (Experimental): Intake of 250 ml of tap water and 100 g of bread baked with 50% gene-modified high-amylose barley and 50% wheat. Consumed over maximum 10 minutes at time 0 min after overnight fasting. At one of four visits.
  The gene-modified barley is produced by researchers at Aarhus and Copenhagen Universities as published in 'Carciofi M, et al., Concerted suppression of all starch branching enzyme genes in barley produces amylose-only starch granules. BMC Plant Biol. 2012 Nov 21;12:223. doi: 10.1186/1471-2229-12-223' The wheat flour is standard commercial available flour.
  Interventions: Dietary Supplement: 50% gene-modified high-amylose barley and 50% wheat

INTERVENTIONS:
Dietary Supplement: 100% wheat — 100 g of bread backed with 100% wheat
  Arms: 100 g of 100% wheat bread
Dietary Supplement: 50% nude barley and 50% wheat — 100 g of bread backed with 50% nude barley and 50% wheat
  Arms: Nude barley 50%
Dietary Supplement: 75% nude barley and 25% wheat — 100 g of bread backed with 75% of nude barley and 25% wheat
  Arms: Nude barley 75%
Dietary Supplement: 50% gene-modified high-amylose barley and 50% wheat — 100 g of bread backed with 50% gene-modified high-amylose barley and 50% wheat
  Arms: Gen-modified high-amylose barley

SUMMARY:
In a series of double-blinded randomized cross-over acute studies, the investigators want to study the effects of different types of barley on the glycemic index (GI) in subjects with type 2 diabetes.

The most common type of barley in Denmark is with rind and demands processing before use. Processing may remove important nutrients from the barley. Some of the original antiquity barley has a loose rind (nude barley), that falls off during harvesting, and thereby reduces the need for processing. The investigators want to study how this ancient type of barley affects GI.

Furthermore, some of the investigators collaborative partners have made it possible to increase the amount of amylose in regular barley by genetic modification. The investigators want to study the effect on GI of this new type of modified barley.

DETAILED DESCRIPTION:
Approx. 60 mio. people worldwide live with diabetes and the prevalence is increasing. The increase is primarily due to obesity, unhealthy diet and lack of physical activity. Therefore, it is important to find dietary products that counteracts this development.

Intake of food with a low glycemic index (GI) reduces the risk of developing type 2 diabetes (T2D) and helps in the regulation of a preexisting diabetes.

Barley has shown some beneficial effects on GI compared with wheat, however, barley is not commonly used in bread making in Denmark.

The most common type of barley in Denmark is with rind and demands processing before use. Processing may remove important nutrients from the barley. Some of the original antiquity barley has a loose rind (nude barley), that falls of during harvesting, and thereby reduces the need for processing. However, it is not known how this ancient type of barley affects GI.

The composition of the starch in barley is of importance when the grain is degraded after consumption. The starch consists of both amylose (which is slowly degraded) and amylopectin (which is quickly degraded). By genetic modification, it was possible for collaborative researchers at the Universities of Aarhus and Copenhagen to increase the amount of amylose in regular barley. Slowly degraded starch is expected to decrease GI.

In a series of acute studies the investigators want to study the effects on the glucose metabolism to intake of bread made with different compositions of wheat, nude barley and gene-modified high-amylose barley in subjects with T2D.

It is expected that both nude barley and gene-modified high-amylose barley lowers the postprandial glycemic response more than wheat and hereby positively affect the glycemic regulation for subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (T2D) defined by standard Danish guidelines.
* HbA1c between 48-78 mmol/l.
* Treatment with drugs for hypertension and high cholesterol is allowed if the treatment dose is stable and does not demand changes during the study period.
* Participants are encouraged to maintain their present psychical activity level and their smoking and alcohol habits.

Exclusion Criteria:

* Type 1 diabetes
* Insulin demanding T2D
* Use of weekly administrated GLP-1 antagonist (e.g. ozempic, trulicity or byetta)
* Use of acarbose
* Significant cardiovascular, kidney, liver or endocrine comorbidity
* Significant psychiatric history
* Treatment with steroids
* Alcohol or drug abuse
* Pregnancy or breastfeeding
* Legally incompetent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemic response | Change from -10 minutes to 240 minutes after bread intake (measured at time -10,0,10,20,30,45,60,90,120,150,180,210,240 minutes)
  Area under the curve for glucose (mmol/L)

SECONDARY OUTCOMES:
Postprandial insulin response | Change from -10 minutes to 240 minutes after bread (measured at time -10,0,10,20,30,45,60,90,120,150,180,210,240 minutes)
  Area under the curve for insulin (pmol/L)
Postprandial glucagon response | Change from -10 minutes to 240 minutes after bread (measured at time -10,0,10,20,30,45,60,90,120,150,180,210,240 minutes)
  Area under the curve for glucagon (pg/mL)
Postprandial triglyceride response | Change from -10 minutes to 240 minutes after bread (measured at time -10,0,30,60,120,180,240 minutes)
  Area under the curve for triglyceride (mmol/L)
Postprandial free fatty acid response | Change from -10 minutes to 240 minutes after bread (measured at time -10,0,30,60,120,180,240 minutes)
  Area under the curve for free fatty acids (mmol/L)
Postprandial GLP-1 (glucagon-like peptide-1) response | Change from -10 minutes to 240 minutes after bread (measured at time -10,0,30,60,120,180,240 minutes)
  Area under the curve for GLP-1 (pmol/L)
Postprandial GIP (Glucose-dependent insulinotropic polypeptide) response | Change from -10 minutes to 240 minutes after bread (measured at time -10,0,30,60,120,180,240 minutes)
  Area under the curve for GIP (pmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Mette B Larsen, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Bohl M, Gregersen S, Zhong Y, Hebelstrup KH, Hermansen K. Beneficial glycaemic effects of high-amylose barley bread compared to wheat bread in type 2 diabetes. Eur J Clin Nutr. 2024 Mar;78(3):243-250. doi: 10.1038/s41430-023-01364-x. Epub 2023 Nov 8. PMID 37940671